CLINICAL TRIAL: NCT00836212
Title: Adjusting Antiretroviral Therapy Dosage Using Therapeutic Drug Monitoring
Acronym: TDM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: Swiss HIV Cohort Study (Network)
Responsible Party: Alexandra Calmy / Doctor, University Hospital, Geneva
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHCS 571
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Human Immunodeficiency Virus; HIV Infections
Keywords: HIV; Adjusting Antiretroviral Therapy; Dosage using Therapeutic Drug Monitoring; Swiss HIV Cohort Study; HIV Geneva; lopinavir; efavirenz; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

ARMS (2):
- LPV (Experimental): Patients with blood levels measured 2 times at 2 weeks intervals in the upper quartile (>percentile 75) of concentrations reported under standard therapy (i.e. EFV 600 mg q.d. or LPV/r 400 or 533 mg bid) will have their dose reduced by approximately one third, with the aim to bring their concentration in the 25-75% percentile range.
  Interventions: Drug: Reducing dose of Lopinavir
- EFV (Experimental): Patients with blood levels measured 2 times at 2 weeks intervals in the upper quartile (>percentile 75) of concentrations reported under standard therapy (i.e. EFV 600 mg q.d. or LPV/r 400 or 533 mg bid) will have their dose reduced by approximately one third, with the aim to bring their concentration in the 25-75% percentile range.
  Interventions: Drug: Reducing dose of efavirenz

INTERVENTIONS:
Drug: Reducing dose of Lopinavir — Patients with blood levels measured 2 times at 2 weeks intervals in the upper quartile (>percentile 75) of concentrations reported under standard therapy (i.e. EFV 600 mg q.d. or LPV/r 400 or 533 mg bid) will have their dose reduced by approximately one third, with the aim to bring their concentration in the 25-75% percentile range.
  Arms: LPV
Drug: Reducing dose of efavirenz — Patients with blood levels measured 2 times at 2 weeks intervals in the upper quartile (>percentile 75) of concentrations reported under standard therapy (i.e. EFV 600 mg q.d. or LPV/r 400 or 533 mg bid) will have their dose reduced by approximately one third, with the aim to bring their concentration in the 25-75% percentile range.
  Arms: EFV

SUMMARY:
Background

Low concentrations of protease inhibitors (PIs) or nonnucleoside reverse transcriptase inhibitors (NNRTIs) are associated with an increased risk of virological failure. Likewise, excessive antiretroviral drug concentrations increase the risk of toxicity. Therapeutic drug monitoring (TDM) may identify and correct excessively high or low PI and/or NNRTI concentrations, and thus minimize toxicity and risk of treatment failure. Treatment guidelines only recommend using TDM to help optimize ARV therapy in selected patients, and there are no clear recommendations to guide the clinician who decides to adjust drug doses. Prospective studies have demonstrated the relationship between EFV plasma concentration and neuropsychiatric symptoms. Moreover, EFV is metabolized mainly by cytochrome P450 2B6 and its concentration was reported to be associated with the CYP2B6 516GrT genetic polymorphism.

For drugs such as EFV or LPV/r, lower doses than the ones validated for standard clinical use have demonstrated efficacy in dose-ranging studies.

The investigators will use a standardised algorithm to reduce doses in patients with plasma EFV or LPV/r concentration above percentile 75. This algorithm is based on a Bayesian approach from the pharmacology unit in Lausanne. The investigators hypothesize that a dosage individualisation is feasible and safe.

2.2 Study Aims

The investigators aim at testing a simplified algorithm for dose reduction in patients with documented virological efficacy, treated by a stable LPV/r or EFV based regimen with elevated plasma concentration of these drugs.

Study Design

Prospective open label study in which all eligible patients screened with a plasma drug concentration of either EFV or LPV/r above percentile 75 will be included. After confirmation of the results at baseline, patients will be offered to decrease drug dosage by a third or a half according to a standardised algorithm. All patients will undergo HIVRNA, biochemistry and validated questionnaires after 3 and 6 months to assess the safety and the benefit of this strategy.

ELIGIBILITY:
Inclusion Criteria:

* Stable regimen including either EFV or LPV/r
* HIVRNA below 40 copies since at least 3 months
* Antiretroviral drug concentration (EFV, LPV/r) plasma concentration at screening above P75
* Signed consent for the SHCS genetics core project

Exclusion Criteria:

* Concomitant medication:Amiodarone, bepidril, flecainide, propafenone, quinidine,Astemizole, terfenadine,Dihydroergotamine, ergotamine,Midazolam, triazolam,Cisapride,Pimozide,Rifabutin
* Renal or hepatic impairment
* Pregnancy or wish to become pregnant within the next 6 months
* Both EFV and LPV/r as part of the antiretroviral drug regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients who reach a plasma concentration within targets (P25-P75) after at least one cycle (and maximum two cycles) of dose reduction according to the provided algorithm at 6 months | 6 months

SECONDARY OUTCOMES:
Number of patients who reach a plasma concentration within targets (P25-P75) after at least one cycle of dose reduction -percentage of spared drugs through TDM-guided dosage adaptation over a 6 months period. Compliance: electronic pills count | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra AC Calmy, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hopistal of Geneva, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- See also: Profil of Alexandra Calmy — http://www.doctorswiss.ch/alexandra-calmy/
- See also: Swiss HIV Cohort Study — http://www.shcs.ch